CLINICAL TRIAL: NCT01794637
Title: Study of Peripheral Microcirculatory Dysfunction in End-stage Liver Disease Patients During Liver Transplantation Using Near Infrared Spectroscopy
Brief Title: Study of Peripheral Tissue Oxygenation in End-stage Liver Disease Patients During Liver Transplantation
Status: Withdrawn | Type: Observational
Why Stopped: Disposables required for the measurements in short supply and not provided by the company / supplier
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Achal Dhir, Principle Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 103363
Record Dates: First submitted 2013-01-17; First posted 2013-02-20 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: End Stage Liver Disease
Keywords: End stage liver disease; Peripheral microcirculatory dysfunction; Liver transplantation; Near infrared spectroscopy
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- the end-stage liver disease patients: the end-stage liver disease scheduled for liver transplantation

SUMMARY:
End - stage liver disease can cause many problems to the patients including fatigue, weakness,jaundice, confusion, abdominal pain and distension. Another important problem is the cardiovascular system (heart and blood vessels). There will be the impairment of heart function to pump blood to the distal part of the body. Blood vessels are also affected by the imbalance of chemical agents which are not detoxified by diseased liver, resulting in impairment of oxygen carrying capacity and tissue oxygen exchange. Mechanism of this process is still poorly understood.

This is a study about the peripheral vascular dysfunction by means of vascular occlusion test (VOT). Blood pressure cuff is inflated (to occlude the proximal vessels and induce distal part ischemia), then deflated and observing the distal tissue oxygenation (StO2)change by the probe (Near-infrared spectroscopy : NIRS) at the hand. From our knowledge, there is no study in patients undergoing liver transplantation.

The study investigator would like to observe the change in peripheral tissue oxygenation in different time points during the liver transplantation. We hypothesize that there is a change in microcirculatory function and StO2 in end-stage liver disease patients detected by VOT and NIRS.

DETAILED DESCRIPTION:
End - stage liver disease patients scheduled for liver transplantation will be enrolled. They will receive normal standard of care. The VOT assessment using a non-invasive, integrated research device (InspectraTM StO2 Vascular Occlusion test (VOT) Research Device Hutchinson Corp Minn, MN, USA) and 15 mm Inspectra thenar sensor probe. An integrated blood pressure cuff is placed on the right arm and inflated to a pressure sufficient to produce arterial inflow occlusion (50mmHg above systolic pressure). The cuff remains inflated until a StO2 value of 40% is achieved. During the inflation and deflation, various StO2 parameters are measured and recorded at designed time point.

Specific VOT parameters of interest:

* Baseline StO2 (reflective of perfusion/metabolism ratio)
* Ischemia slope (partly reflective of basal O2 consumption)
* Ischemia area (partly reflective of basal O2 consumption)
* Time till 40% ischemic threshold (partly reflective of basal O2 consumption)
* Recovery slope (biphasic and reflective of shear stress and endothelial vasoreactivity)
* Recovery area (reflective of endothelial vasoreactivity)
* Hyperemia area (reflective of endothelial vasoreactivity and tissue metabolic rate) To determine effect of core versus peripheral temperatures, a conventional skin thermocouple will be placed under adhesive patch used to secure NIRS optodes in position on thenar eminence

Data collection

1. Demographic data: a)age, b)sex, c)diagnosis, d)Model of End-stage Liver Disease (MELD) score, Body Mass Index (BMI)
2. Clinical parameter : the investigator will collect clinical data including VOT parameters (from above), hemodynamics parameter, chemical parameters and medications used in specific time frame :

   * time frame

     1. pre-operative (for base line data)
     2. pre-anhepatic phase (15 min. before the inferior vena cava (IVC) clamps)
     3. anhepatic phase (30 min. after the IVC clamps),
     4. reperfusion phase (30 min. after the release the IVC clamps),
     5. immediately post operation (at the skin closure)
   * hemodynamics : SpO2 (Pulse oxygen saturation), MAP (mean arterial pressure), HR (heart rate), CVP (Central venous pressure), PAP (Pulmonary artery pressure), CI (Cardiac output index), PCWP (Pulmonary artery wedge pressure), SVRI (Systemic vascular resistance index), PVRI (Pulmonary vascular resistance index), temperature
   * chemical : Hb, Platelets, INR (international normalized ratio) (PT : Prothrombin time), PTT (partial thromboplastin time), Lactate, base excess
   * Medications : Volatile agents, Vasopressors (Concentration at recorded time points)

Then we will compare the dynamic changes of StO2 parameters in different time points (as mentioned) and compare to the hemodynamics and chemical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients suffering from end-stage liver disease scheduled for liver transplantation.

Exclusion Criteria:

* Patients with known peripheral vascular disease
* Patients receiving Oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients suffering from end-stage liver disease scheduled for liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
the significant changes in StO2 between anhepatic and reperfusion phase of the end-stage liver disease patient undergoing liver transplantation | compare the change of StO2 during different phase of the liver transplantation (base line, pre-anhepatic phase, anhepatic phase, re-perfusion phase and at skin closure)
  Our data measured will be included only during the operation and at skin closure can reflect early postoperative period.

SECONDARY OUTCOMES:
dynamic changes in StO2 during liver transplantation with possible correlation with hemodynamic or chemical parameters in different time points | preoperative for baseline data, intraoperative (during different phase of liver transplantation) and finish data record at skin closure time)
  from previous study indicates that new liver start its metabolic function well right after the vascular connection complete. So, the investigator want to analyze the correlation between the dynamic StO2 changes during operative period

CONTACTS AND LOCATIONS:
Overall Officials: Achal Dhir, MD, Principal Investigator — Western University
Locations (1):
- University Hospital, London Health Science Center, London, Ontario, Canada

REFERENCES:
- [Background] Groszmann RJ. Hyperdynamic circulation of liver disease 40 years later: pathophysiology and clinical consequences. Hepatology. 1994 Nov;20(5):1359-63. No abstract available. PMID 7927273
- [Background] Helmy A, Newby DE, Jalan R, Johnston NR, Hayes PC, Webb DJ. Nitric oxide mediates the reduced vasoconstrictor response to angiotensin II in patients with preascitic cirrhosis. J Hepatol. 2003 Jan;38(1):44-50. doi: 10.1016/s0168-8278(02)00319-7. PMID 12480559
- [Background] Okumura H, Aramaki T, Katsuta Y, Terada H, Satomura K, Akaike M, Sekiyama T. Regional differences in peripheral circulation between upper and lower extremity in patients with cirrhosis. Scand J Gastroenterol. 1990 Sep;25(9):883-9. doi: 10.3109/00365529008997608. PMID 2218394
- [Background] Caraceni P, Dazzani F, Salizzoni E, Domenicali M, Zambruni A, Trevisani F, Bernardi M. Muscle circulation contributes to hyperdynamic circulatory syndrome in advanced cirrhosis. J Hepatol. 2008 Apr;48(4):559-66. doi: 10.1016/j.jhep.2007.12.016. Epub 2008 Jan 31. PMID 18276031
- [Background] Seino Y, Ohki K, Nakamura T, Tsukamoto H, Takano T, Aramaki T, Okumura H, Hayakawa H. Pathophysiological characteristics of cutaneous microcirculation in patients with liver cirrhosis: relationships to cardiovascular hemodynamics and plasma neurohormonal factors. Microvasc Res. 1993 Sep;46(2):206-15. doi: 10.1006/mvre.1993.1047. PMID 8246819
- [Background] Poeze M. Tissue-oxygenation assessment using near-infrared spectroscopy during severe sepsis: confounding effects of tissue edema on StO2 values. Intensive Care Med. 2006 May;32(5):788-9. doi: 10.1007/s00134-006-0121-x. Epub 2006 Mar 17. No abstract available. PMID 16544119
- [Background] Harel F, Denault A, Ngo Q, Dupuis J, Khairy P. Near-infrared spectroscopy to monitor peripheral blood flow perfusion. J Clin Monit Comput. 2008 Feb;22(1):37-43. doi: 10.1007/s10877-007-9105-9. Epub 2007 Nov 27. PMID 18040873
- [Background] Thomson SJ, Cowan ML, Forton DM, Clark SJ, Musa S, Grounds M, Rahman TM. A study of muscle tissue oxygenation and peripheral microcirculatory dysfunction in cirrhosis using near infrared spectroscopy. Liver Int. 2010 Mar;30(3):463-71. doi: 10.1111/j.1478-3231.2009.02157.x. Epub 2009 Nov 16. PMID 19912533
- [Background] Steib A, Freys G, Gohard R, Curzola U, Ravanello J, Lutun P, Boudjema K, Otteni JC. Tissue oxygenation during liver transplantation. Crit Care Med. 1992 Jul;20(7):977-83. doi: 10.1097/00003246-199207000-00013. PMID 1617992
- [Background] Al-Hamoudi WK, Alqahtani S, Tandon P, Ma M, Lee SS. Hemodynamics in the immediate post-transplantation period in alcoholic and viral cirrhosis. World J Gastroenterol. 2010 Feb 7;16(5):608-12. doi: 10.3748/wjg.v16.i5.608. PMID 20128030
- [Background] Shelly MP, Dixon JS, Park GR. The pharmacokinetics of midazolam following orthotopic liver transplantation. Br J Clin Pharmacol. 1989 May;27(5):629-33. doi: 10.1111/j.1365-2125.1989.tb03428.x. PMID 2667599
- [Background] Hickman PE, Potter JM, Pesce AJ. Clinical chemistry and post-liver-transplant monitoring. Clin Chem. 1997 Aug;43(8 Pt 2):1546-54. PMID 9265907